CLINICAL TRIAL: NCT05616481
Title: Laparoscopic Burch Colposuspension Versus Modified Burch Colposuspension For Treatment Of Female Stress Urinary Incontinence; Randomized Controlled Trial
Brief Title: Laparoscopic Burch Colposuspension Versus Modified Burch Colposuspension
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Mohamed Fawzy Abd Elfattah Salman, Director, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Burch versus Modefied Burch
Record Dates: First submitted 2022-11-07; First posted 2022-11-15 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Stress Urinary Incontinence; Burch Colposuspention
Keywords: Stress urinary incontinence; Burch Colposuspension; TOT
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic Burch (Active Comparator): The original procedure will be performed
  Interventions: Procedure: Laparoscopic Burch colposuspension
- Laparoscopic modefied Burch procedur (TOT-like) (Active Comparator): Sutures on the pubocervical fascia are placed at the level of the attachment of the arcus tendinous fascia pelvis and the pubourethral ligament.
  Interventions: Procedure: Modefied Burch (TOT - like)

INTERVENTIONS:
Procedure: Laparoscopic Burch colposuspension — The original Burch procedure will be performed
  Arms: Laparoscopic Burch
Procedure: Modefied Burch (TOT - like) — more lateral fixation to avoid post-operative voiding dysfunction
  Arms: Laparoscopic modefied Burch procedur (TOT-like)

SUMMARY:
This study aims to compare the success rate and complications following laparoscopic standard Burch colposuspension and laparoscopic modified Burch colposuspension (Transobturator tape like)

ELIGIBILITY:
Inclusion Criteria:

* Women with genuine stress urinary incontinence.
* Mixed urinary incontinence with predominant stress element.
* Refractory cases to conservative therapy or patients who are not willing to consider (further) conservative treatment.

Exclusion Criteria:

* Mixed incontinence with predominant Urge urinary incontinence.
* Recent pelvic surgery (less than 3 months).
* Neurogenic lower urinary tract dysfunction.
* Previous surgery for stress urinary incontinence.
* Pregnancy
* Less than 12 months post-partum.
* Other gynaecologic pathologies affecting bladder functions ( eg, fibroids, ovarian cysts)
* Genito-urinary malignancy.
* Current chemo or radiation therapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
The success rates of both laparoscopic Burch colposuspension versus laparoscopic modified Burch colposuspension for treatment of female stress urinary incontinence | 3 months post operative

SECONDARY OUTCOMES:
Post operative rates of voiding dysfunction (at 3 months). | at 3 months
Overall operative time | Intraoperative (measured from verrus needle insertion)
Complication rates of both techniques. | up to 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Fawzy Salman, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Abrar S, Razzak L, Mohsin R. The practice of Burch Colposuspension versus Mid Urethral Slings for the treatment of Stress Urinary Incontinence in developing country. Pak J Med Sci. 2021 Sep-Oct;37(5):1359-1364. doi: 10.12669/pjms.37.5.4017. PMID 34475912
- [Background] Aleksandrov A, Meshulam M, Rabischong B, Botchorishvili R. Laparoscopic TOT-like Burch Colposuspension: Back to the Future? J Minim Invasive Gynecol. 2021 Jan;28(1):24-25. doi: 10.1016/j.jmig.2020.04.018. Epub 2020 Apr 24. PMID 32339752
- [Background] Carmel ME, Deng DY, Greenwell TJ, Zimmern PE. Definition of Success after Surgery for Female Stress Incontinence or Voiding Dysfunction: An Attempt at Standardization. Eur Urol Focus. 2016 Aug;2(3):231-237. doi: 10.1016/j.euf.2016.03.005. Epub 2016 Mar 26. PMID 28723368
- [Background] Kim A, Kim S, Kim HG. Current Overview of Surgical Options for Female Stress Urinary Incontinence. Int Neurourol J. 2020 Sep;24(3):222-230. doi: 10.5213/inj.2040052.026. Epub 2020 Sep 30. PMID 33017893
- [Background] Marquini GV, Bella ZIKJD, Sartori MGF. Burch Procedure: A Historical Perspective. Rev Bras Ginecol Obstet. 2022 May;44(5):511-518. doi: 10.1055/s-0042-1744312. Epub 2022 Feb 18. PMID 35181882